CLINICAL TRIAL: NCT00630656
Title: A Phase 2 Randomized, Double-blind, Placebo-controlled Study of the Safety and Efficacy of Talactoferrin Alfa in Patients With Severe Sepsis
Brief Title: Safety and Efficacy Study of Recombinant Human Lactoferrin to Treat Severe Sepsis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Agennix (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LF-0801; NIH grant 1R44GM077816-01A2
Record Dates: First submitted 2008-02-28; First posted 2008-03-07 (Estimated); Last update posted 2011-08-23 (Estimated); Status verified 2011-08

CONDITIONS: Severe Sepsis
Keywords: sepsis; talactoferrin; lactoferrin; recombinant human lactoferrin
MeSH Terms: conditions — Sepsis | interventions — talactoferrin alfa

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Talactoferrin alfa
  Interventions: Drug: Talactoferrin alfa
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Talactoferrin alfa — 15 mL of an oral solution of 100mg/mL (1.5 g) given 3 times a day for up to 28 days or until discharge from the intensive care unit
  Arms: 1
Drug: Placebo — Placebo given 3 times a day for up to 28 days or until discharge from the intensive care unit
  Arms: 2

SUMMARY:
Study will evaluate the safety and potential benefit of recombinant human talactoferrin as an addition to the standard care of severe sepsis.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* Onset of severe sepsis within the previous 24 hours
* Must be receiving antibiotic therapy
* Informed consent form signed by patient, legal next-of-kin or legal guardian
* Able to take medication by mouth or feeding tube

Exclusion Criteria:

* Receipt of investigational medication within 4 weeks prior to participation in the study
* Pregnant or breast-feeding
* Severe congestive heart failure
* Known severe HIV infection
* Presence of severe burns
* Patients on high dose immunosuppressants
* Patients whose death is considered imminent
* Patients whose life expectancy for concurrent illness is less than 6 months
* Severe hypoxic encephalopathy or persistent vegetative state
* Severe liver disease
* Patient, legal representative or patient's primary physician not committed to providing full, aggressive life support

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2008-04; Primary Completion 2009-08 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | 28-day

SECONDARY OUTCOMES:
All-cause mortality | 3 months
All-cause mortality | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Kalpalatha K Guntupalli, MD, Principal Investigator — Baylor College of Medicine
Locations (34):
- United States (27):
  - Loma Linda University Medical Center, Loma Linda, California
  - UC Davis Medical Center, Sacramento, California
  - Olive View- UCLA Medical Center, Sylmar, California
  - Denver Health Medical Center, Denver, Colorado
  - The George Washington University Hospital, Washington D.C., District of Columbia
  - Rush University Medical Center, Chicago, Illinois
  - West Suburban Medical Center, Oak Park, Illinois
  - Floyd Memorial Hospital and Health Services, New Albany, Indiana
  - University of Iowa Hospitals and Clinic, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Baystate Medical Center, Springfield, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - St. Louis University, St Louis, Missouri
  - St. John's Mercy Medical Center, St Louis, Missouri
  - Cooper University Hospital, Camden, New Jersey
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Oklahoma Health Science Center, Oklahoma City, Oklahoma
  - University of Pittsburgh Medical Center Presbyterian Hospital, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Texas Tech University Health Sciences Center, El Paso, Texas
  - Ben Taub General Hospital, Houston, Texas
  - The Methodist Hospital, Houston, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Scott & White Memorial Hospital, Temple, Texas
  - Intermountain Medical Center, Salt Lake City, Utah
- Canada (2):
  - Vancouver General Hospital, Vancouver, British Columbia
  - Kingston General Hospital, Kingston, Ontario
- France (2):
  - Centre Hospitalier de Montauban, Montauban
  - Centre Hospitalier Angouleme, Saint-Michel
- Helios Klinikum Erfurt, Erfurt, Germany
- Spain (2):
  - Hospital de Sabadell, Sabadell, Catalonia
  - Hospital Mutua de Terrassa, Terrassa, Catalonia

REFERENCES:
- [Derived] Guntupalli K, Dean N, Morris PE, Bandi V, Margolis B, Rivers E, Levy M, Lodato RF, Ismail PM, Reese A, Schaumberg JP, Malik R, Dellinger RP; TLF LF-0801 Investigator Group. A phase 2 randomized, double-blind, placebo-controlled study of the safety and efficacy of talactoferrin in patients with severe sepsis. Crit Care Med. 2013 Mar;41(3):706-16. doi: 10.1097/CCM.0b013e3182741551. PMID 23425819